CLINICAL TRIAL: NCT06267469
Title: Boutonniere Deformity Effectiveness of Thermoplastic and Fabricated Orthoses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magdalena Kolasińska (Other)
Collaborators: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Responsible Party: Sponsor-Investigator, Magdalena Kolasińska, Principal Investigator, Józef Piłsudski University of Physical Education
Organization: Józef Piłsudski University of Physical Education (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Boutonniere deformity
Record Dates: First submitted 2024-02-03; First posted 2024-02-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Orthotic Devices
Keywords: Boutonniere deformity; thermoplastic orthosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Grip strength (Other): Using a hydraulic handgrip dynamometer by Saehan according to the procedure to measure grip strength
  Interventions: Device: Thermoplastic orthosis
- DASH Questionnaire (Other): The DASH questionnaire assesses upper limb disability and consists of 30 questions in the general section and an additional work module with 4 questions and a sport/instrument playing module with 4 questions. Assess symptoms and the inability to perform certain activities based on health status.
  Interventions: Device: Thermoplastic orthosis
- Likert scale (Other): Measurement strategy, used in surveys to gain knowledge about the degree of acceptance of the orthosis
  Interventions: Device: Thermoplastic orthosis
- Kapandji score (Other): Is a tool useful for assessing the opposition of the thumb
  Interventions: Device: Thermoplastic orthosis
- NRS scale (Other): Requires the patient to rate their pain on a defined scale
  Interventions: Device: Thermoplastic orthosis
- Pinch strength (Other): Using a hydraulic handgrip dynamometer by Saehan according to the procedure to measure grip strength
  Interventions: Device: Thermoplastic orthosis

INTERVENTIONS:
Device: Thermoplastic orthosis — The use of the author's orthosis is aimed at correcting the anatomical alignment of the MP (metacarpophalangeal) joints, IP (interphalangeal) by properly tensioning the central extensor band and the lateral bands of the thumb's extensor apparatus. It should significantly increase the mobility of the hand in connection with improving hand grip and reducing pain.

SUMMARY:
The goal of this study is to present the author's thumb orthosis with a butonier deformity and its effect on hand function, strength, dexterity and pain levels in relation to patients wearing factory-made orthopedic supplies. It is planned to include about 60 people in the study (30 people each in the group with thermoplastic orthoses and 30 participants with factory-made orthoses)

The main questions it aims to answer are:

1. How much improvement in dexterity will the patient wearing the orthosis get? 2. By how much will the grip strength of the whole hand and pincer grip strength improve with the orthosis? 3. How will wearing the orthosis affect the pain associated with the disease? Participants will

1. measurement of grip strength of the right and left hands with a dynamometer in an orthosis and without an orthosis, at the time of the test conducted and at the appointed times.
2. measurement of pincer grip strength with a dynamometer in an orthosis and without an orthosis, at the time of the test conducted and at the designated times.

4. completion of the DASH questionnaire 6. assessment of the NRS pain scale in relation to the period of 6 months before the start of the study 7. Likert scale - evaluation of satisfaction with the use of the orthosis 8. the Kapandji scale Researchers will compare patients with thermoplastic orthosis and patients with fabric orthosis to see which is more functional.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with RA
* diagnosed thumb deformity: butonier finger, type I or II
* female
* age 18 - 65 years
* patient's consent to the study

Exclusion Criteria:

* other deformity of the thumb
* less than 1 year since surgical intervention in the hand
* less than 6 months since delivery injections within the thumb
* change in treatment during the study and 3 months before the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Grip strength | 6 month
  Measurement of grip strength and of the right and left hands with a dynamometer in an orthosis and without an orthosis.
DASH -Disabilities of the Arm, Shoulder and Hand | 6 month
  The DASH questionnaire assesses upper limb disability and consists of 30 questions in the general section and an additional work module with 4 questions and a sport/instrument playing module with 4 questions. In the DASH a higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. The score on test ranges from 0 (no disability) to 100 (most severe disability)
Likert scale | 6 month
  Measurement strategy, used surveys through which knowledge about the degree of acceptance of the product can be obtained. Participants provide data using a four-point strongly disagree, disagree, agree, strongly agree
Kapandji score | 6 month
  Is a tool useful for assessing the opposition of the thumb. A score of 0 indicates no opposition, a score of 10 indicates maximal opposition.
NRS - Numerical Rating Scale | 6 month
  Requires the patient to rate their pain on a defined scale. Ranges from 0 to 10. zero being an example of someone with no pain and ten being the worst pain possible.
pinch strength | 6 month
  pincer grip strength of the right and left hands with a dynamometer in an orthosis and without an orthosis.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Kolasińska, Msc, Study Director — University of Physical Education in Warsaw
Locations (2):
- Poland (2):
  - Terapia Ręki Magda Kolasińska, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. prof. dr hab. med. Eleonory Reicher, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: No